CLINICAL TRIAL: NCT01264263
Title: Prevalence of Subclinical Atherosclerosis and Its Associated Factors in Hyperlipidemic Korean Adults With Diabetes
Acronym: ALTO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CKR-DUM-2010/1
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus; Dyslipidemia
Keywords: cIMT; hs CRP (C-reactive protein); DM (Diabetic Mellitus); Korea; Corelation between cIMT (carotid intima media thickness); Cardio Vascular risk in Diabetic Mellitus
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood and serum, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study is to investigate correlation between Carotid Intima Media Thickness (cIMT) and several factors such as; hs C-reactive protein (CRP), HbA1c, lipid profile in Korean diabetic patients with atherosclerosis. Total 360 patients will be enrolled through 6 sites.

DETAILED DESCRIPTION:
MC MD

ELIGIBILITY:
Inclusion Criteria:

* patients with Diabetic Mellitus
* patients with dyslipidemia

Exclusion Criteria:

* patients who have established cardiovascular disease
* patient using NSAID

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 360 patients who has diabetic mellitus with dyslipidemia
Sampling Method: Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measurement of intima media thickness, visit 1 | Visit 1
Measurement of intima media thickness, visit 2 | Visit 2

SECONDARY OUTCOMES:
hs-C-Reactive Protein, visit 1 | Visit 1
hs-C-Reactive Protein, visit 2 | Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Dongsun Kim, Study Chair — Hanyang University; Eunkyung Hong, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital; Hyunsang Kwon, Principal Investigator — Yeoido Saint Mary's Hospital; Dongjoon Kim, Principal Investigator — Ilsan-Paik Hospital; Sungjin Lee, Principal Investigator — Hallym University Hospital; Singon Kim, Principal Investigator — Korea University Anam Hospital
Locations (3):
- South Korea (3):
  - Research Site, Anyang
  - Research Site, Koyang
  - Research Site, Seoul

REFERENCES:
- [Derived] Hong EG, Ohn JH, Lee SJ, Kwon HS, Kim SG, Kim DJ, Kim DS. Clinical implications of carotid artery intima media thickness assessment on cardiovascular risk stratification in hyperlipidemic Korean adults with diabetes: the ALTO study. BMC Cardiovasc Disord. 2015 Oct 6;15:114. doi: 10.1186/s12872-015-0109-y. PMID 26438201